CLINICAL TRIAL: NCT05638607
Title: Effect of Intensified Occupational Therapy on Basic Activities of Daily Living: a Randomized Controlled Trial
Brief Title: Effect of Intensified Occupational Therapy on Basic Activities of Daily Living
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1-10-72-169-22
Record Dates: First submitted 2022-11-14; First posted 2022-12-06 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: ADL
Keywords: Stroke; Occupational therapy; Trial; Basic activities of daily living
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensified occupational therapy (Experimental): Two hours occupational therapy each weekday with specific focus on basic ADL
  Interventions: Behavioral: Intensified occupational therapy
- Usual care (Active Comparator): Occupational therapist instruct nursing staff on how to assist patients with basic ADL
  Interventions: Behavioral: Intensified occupational therapy

INTERVENTIONS:
Behavioral: Intensified occupational therapy — The intervention is an intensified occupational therapy effort, which does not take time away from other occupational therapy efforts.

SUMMARY:
The objective is to investigate the effect of an intensified occupational therapy intervention on independence in basic activities of daily living (ADL) in subjects with stroke

ELIGIBILITY:
Inclusion Criteria:

* First-time stroke
* <=4 on four of six Functional Independence Measure (FIM) basic ADL items

Exclusion Criteria:

* Not able to understand danish

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Assessment of motor and process skills (AMPS) | Change in scores from baseline to scores following three weeks intervention
  Observed limitations in activities of daily living, with scores for the motor- and proces- domains of activitites of daily living abilities. Each item in the domains is scored on a 4-point Likert scale, with higher scores representing a better outcome.

SECONDARY OUTCOMES:
Activities of Daily Living - Interview | Change in scores from baseline to scores following three weeks intervention
  Patient reported outcome measure
Functional Independence Measure (FIM) | Change in scores from baseline to scores following three weeks intervention
  FIM measures activities of daily living observed by the interdisciplinary team in routinely daily practice. The scale has 18 items which are scored on a 7 point Likert Scale. The total score thus range from 18 to 126, with higher scores represent a better outcome.
Goal Attainment Scaling | Following three weeks intervention
  Scoring system based on rehabilitation goal setting. Each rehabilitation goal is rated on a 5-point Likert scale from -2 to +2 with higher score representing a better outcome. Examples are: -2 denoting "much less than expected" and +2 denoting "much more than expected".
Length of stay | Follow-up up to one year of admission for inpatient rehabilitation.
  Length of stay starts the day the patient is admitted for subacute rehabilitation and ends the day the patient is discharged. The mean length of stay at the hospital is arround 6 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Fabricius, PhD, Principal Investigator — Hammel Neurorehabilitation Centre and University Research Clinic
Locations (1):
- Hammel Neurorehabilitation Centre and University Research Clinic, Hammel, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No